CLINICAL TRIAL: NCT06349382
Title: Preoperative Oral Carbohydrate Loading in Aortic Surgery
Brief Title: CArbohydrate Loading in Aortic Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Belgrade (Other)
Responsible Party: Principal Investigator, Igor Koncar, Vascular surgeon, MD, Ph.D., University of Belgrade
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CALAS
Record Dates: First submitted 2024-03-23; First posted 2024-04-05 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Abdominal Aortic Aneurysm; Leriche Syndrome
MeSH Terms: conditions — Aortic Aneurysm, Abdominal; Leriche Syndrome

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to receive preoperative OCHL (the experimental group) or no intervention (the control group) in a 1:1 ratio. Randomization will be performed using computer-generated randomization codes, which will be held in sealed envelopes. Patients in the experimental group (OCHL group) will receive a high-carbohydrate beverage (12.6% carbohydrates, 50 kcal/100 mL, 285 mOsm/kg; PreOp®, Nutricia, Zoetermeer, The Netherlands) 800 mL on the evening before surgery (between 9 p.m. and 11 p.m.), and 400 mL 2 hours before the induction of anesthesia. Participants in the no-intervention (control) group will be fasted from midnight until surgery. All other aspects of perioperative patient care will be the same for all participants, as per the standardized Institutional protocol for the treatment of abdominal aortic aneurysms and Leriche Syndrome.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- OCHL group (Experimental): Approximately 25 patients will receive a high-carbohydrate beverage in the evening before surgery and two hours before the induction of anesthesia.
  Intervention: carbohydrate-rich beverage
  Glucose and insulin values will be assessed from the peripheral venous or arterial blood samples (from the arterial cannula postoperatively), taken at four-time points. Other parameters of insulin resistance (HOMA-IR, HOMA-ISI, and HOMA-β) will be calculated based on the values of fasting insulin and fasting glucose for each of four time points.
  The subjective well-being variables will be evaluated in the morning before the surgery, 6-12 hours after the surgery, and 24 hours after the surgery.
  Interventions: Dietary Supplement: carbohydrate-rich beverage
- Control group (No Intervention): Approximately 25 patients in the no-intervention (control) group will be fasted from midnight until surgery.
  Glucose and insulin values will be assessed from the peripheral venous or arterial blood samples (from the arterial cannula postoperatively), taken at four-time points. Other parameters of insulin resistance (HOMA-IR, HOMA-ISI, and HOMA-β) will be calculated based on the values of fasting insulin and fasting glucose for each of four time points.
  The subjective well-being variables will be evaluated in the morning before the surgery, 6-12 hours after the surgery, and 24 hours after the surgery.

INTERVENTIONS:
Dietary Supplement: carbohydrate-rich beverage — Patients in the OCHL group will drink a high-carbohydrate beverage (12.6% carbohydrates, 50 kcal/100 mL, 285 mOsm/kg; PreOp®, Nutricia, Zoetermeer, The Netherlands) 800 mL in the evening before surgery (between 9 p.m. and 11 p.m.), and 400 mL two hours before the induction of anesthesia.
  Other Names: the experimental group
  Arms: OCHL group

SUMMARY:
The adverse effects of overnight fasting before surgery have been well-documented in the contemporary literature. Still, due to the possibility of pulmonary aspiration of gastric contents, many clinicians worldwide still employ this practice. On the other hand, the benefits of preoperative oral carbohydrate loading (OCHL) have been shown in various patient groups. Studies examining the usefulness of preoperative OCHL in aortic surgery are lacking. In particular, no randomized control trials have specifically examined the impact of preoperative OCHL on the postoperative course in patients undergoing open abdominal aortic surgery.

DETAILED DESCRIPTION:
The aims of the study are: 1) to assess the effect of preoperative OCHL on the postoperative course in terms of length of ICU stay, the incidence of surgical and non-surgical complications, postoperative local wound infections, and short-term (30-days) mortality rate; 2) to evaluate the impact of preoperative OCHL on glucose homeostasis, insulin resistance, and patients' subjective well-being; 3) to compare the differences between preoperative OCHL and a conventional fasting protocol.

A prospective, single-center randomized control trial will include approximately 50 consecutive patients undergoing elective open repair due to abdominal aortic aneurysm or Leriche Syndrome. All patients will be operated on under the conditions of general anesthesia during the period from April to October 2024 at the investigators' Institution.

Basic demographic, anthropometric, and clinical data of interest (data on current disease, comorbidities, smoking status, preoperative chronic therapy, previous operations, and basic laboratory and coagulation parameters) will be collected through patient interviews and obtained from medical records. Data regarding intraoperative and postoperative course (including length of ICU stay, postoperative complications, and intrahospital mortality) will be extracted from medical records and database included in daily practice. Data regarding short-term (30 days) morbidity and mortality will be obtained through telephone interviews or personally - on the postoperative control examinations.

Glucose and insulin values will be assessed from the peripheral venous or arterial blood samples (from the arterial cannula postoperatively), taken at T1, 9-11 p.m. in the evening before the surgery (before high-carbohydrate beverage in OCHL group), T2 90 min after high-carbohydrate beverage ingestion in OCHL group, i.e., at 06 a.m. in the control group, on the day of the surgery, T3 six hours following the surgery, and T4 06 a.m. on the first postoperative day. Other parameters of insulin resistance (Homeostatic Model Assessment for Insulin Resistance, HOMA-IR; insulin sensitivity index, HOMA-ISI; and homeostasis model assessment of β-cell function, HOMA-β) will be calculated based on the following equations: HOMA-IR = [fasting insulin (μU/mL) × fasting glucose (mmol/L)]/22.5; HOMA-ISI = 1/log/[fasting glucose (mmol/L) + fasting insulin (μU/mL)], HOMA-β = (20 × fasting plasma insulin [µU/ml])/(fasting plasma glucose [mmol/L] - 3.5), for each of four-time points. No intravenous fluid administration will be given preoperatively, while intraoperatively, no glucose-containing fluids nor insulin will be administered. Also, patients will not receive intravenous or oral glucose solutions six hours before the postoperative morning blood sampling (from midnight to 06 h). Subjective well-being will be assessed using the visual analog scale (VAS) for the six following aspects: anxiety, hunger, thirst, tiredness, pain, and headache. The patients will be instructed to mark a vertical line on a 100 mm horizontal scale, which will be marked with "no symptom" at its left end (score of zero) and with "the worst possible symptom" (score of 10) at its right end. The distance from the left end to the patient's mark will represent the score of the perceived symptom. The variables of subjective well-being will be evaluated at several time points: in the morning before the surgery, 6-12 hours after the surgery, and 24 hours after the surgery. Local wound infection will be defined as redness, pain, and/or drainage on the surgical site, along with an increase in infectious parameters, with or without fever > 38°C.

A median stay of three days with a standard deviation of one day was noted by analyzing the ICU length of stay in a historical cohort of patients who underwent open elective aortic surgery. A power calculation showed that a total sample size of 32 patients is sufficient to have an 80% chance of detecting, as significant at the 5% level, a decrease in the ICU length of stay from 3 in the control group to 2 days in the experimental group. To allow for dropout, the investigators will recruit 50 patients.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive patients admitted due to elective surgical treatment of abdominal aortic aneurism or Leriche Syndrome.
* Patients scheduled to be operated on first on a given day, that is, patients whose surgery will be performed first in the morning.
* Personally signed informed consent.

Exclusion Criteria:

* Patients with diabetes or fasting glucose level above seven mmol/L;
* Patients with disorders that prolong gastric emptying (gastroesophageal reflux disease, history of gastrointestinal surgery, hiatus hernia or intestinal obstruction);
* Patients with conditions that could potentially prolong the postoperative recovery (severe physical disability, cognitive impairment, autoimmune diseases, severe infection, significant liver and renal failure, or severe psychiatric/mental disorders);
* Patients with alcohol/drug abuse
* Obese patients with obesity class 3 (BMI ≥ 40 kg/m2);
* Patients undergoing emergent surgery;
* Patients treated with immunosuppressants and/or steroids in the past three months before surgery;
* Patients in whom difficult airway is anticipated.

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2024-08-01 (Actual); Primary Completion 2025-02-01 (Actual); Study Completion 2025-04-01 (Actual)

PRIMARY OUTCOMES:
The ICU length of stay | up to 10 days following surgery
  The ICU length of stay will be defined as the interval from the end of surgery to the date of ICU discharge.
Homeostatic Model Assessment for Insulin Resistance (HOMA-IR) | 1 day preoperatively - 1 day following surgery
  Values of glucose and serum insulin will be assessed at four time-points: T1, 9-11 p.m. in the evening before the surgery (before high-carbohydrate beverage in OCHL group); T2 90 min after high-carbohydrate beverage ingestion in OCHL group, i.e., at 06 a.m. in the control group, on the day of the surgery; T3 6 h following the surgery, and T4 06 a.m. on the postoperative day 1. Values of HOMA-IR will be subsequently calculated for each of the four time points.
Insulin sensitivity index (HOMA-ISI) | 1 day preoperatively - 1 day following surgery
  Values of glucose and serum insulin will be assessed at four time-points: T1, 9-11 p.m. in the evening before the surgery (before high-carbohydrate beverage in OCHL group); T2 90 min after high-carbohydrate beverage ingestion in OCHL group, i.e. at 06 a.m. in the control group, on the day of the surgery; T3 6 h following the surgery, and T4 06 a.m. on the postoperative day 1. Values of HOMA-ISI will be subsequently calculated for each of the four time points.
Homeostasis model assessment of β-cell function (HOMA-β) | 1 day preoperatively - 1 day following surgery
  Values of glucose and serum insulin will be assessed at four time-points: T1, 9-11 p.m. in the evening before the surgery (before high-carbohydrate beverage in OCHL group); T2 90 min after high-carbohydrate beverage ingestion in OCHL group, i.e. at 06 a.m. in the control group, on the day of the surgery; T3 6 h following the surgery, and T4 06 a.m. on the postoperative day 1. Values of HOMA-β will be subsequently calculated for each of the four time points.
Six aspects of subjective well-being according to the visual analog scale | preoperatively - 1 day following surgery
  The variables of the subjective well-being will be evaluated in several time points: in the morning before the surgery, 6-12h following the surgery and 24h following the surgery. The minimum score is zero, and the maximum score is 10. The higher the score, the worse the outcome.

SECONDARY OUTCOMES:
Length of hospital stay | From the date of hospital admission until the date of hospital discharge or date of death from any cause, whichever came first, assessed up to two months following surgery.
  Length of hospital stay will be defined as the interval from the admission to the hospital to the date of hospital discharge.
30-day mortality rate | 30 days following surgery
  30-day mortality would refer to any lethal outcome (due to any cause), that would occur 30 days following surgery.
The incidence of local wound infections | 30 days following surgery
  Local wound infection will be defined as redness, pain and/or drainage on the surgical site, along with an increase in infectious parameters, with or without fever > 38°C.
The incidence of postoperative surgical complications | 30 days following surgery
  Postoperative surgical complications will be defined as complications related to the surgical procedure within 30 days after the operation.
The incidence of postoperative non-surgical complications | 30 days following surgery
  Postoperative non-surgical complications will be defined as complications which are not related to surgical procedures/techniques.

CONTACTS AND LOCATIONS:
Overall Officials: Slobodan Cvetkovic, MD, Ph.D., Study Chair — Clinic for Vascular and Endovascular Surgery, University Clinical Center of Serbia
Locations (1):
- Clinic for Vascular and Endovascular Surgery, University Clinical Center of Serbia, Belgrade, Serbia, Serbia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sun J, Wei G, Hu L, Liu C, Ding Z. Perioperative pulmonary aspiration and regurgitation without aspiration in adults: a retrospective observational study of 166,491 anesthesia records. Ann Palliat Med. 2021 Apr;10(4):4037-4046. doi: 10.21037/apm-20-2382. Epub 2021 Mar 23. PMID 33832306
- [Background] Xu D, Zhu X, Xu Y, Zhang L. Shortened preoperative fasting for prevention of complications associated with laparoscopic cholecystectomy: a meta-analysis. J Int Med Res. 2017 Feb;45(1):22-37. doi: 10.1177/0300060516676411. Epub 2017 Jan 12. PMID 28222625
- [Background] Zhou G, Zhu F, An Y, Qin L, Lv J, Zhao X, Shen J. Prolonged preoperative fasting and prognosis in critically ill gastrointestinal surgery patients. Asia Pac J Clin Nutr. 2020;29(1):41-47. doi: 10.6133/apjcn.202003_29(1).0006. PMID 32229440
- [Background] Smith I, Kranke P, Murat I, Smith A, O'Sullivan G, Soreide E, Spies C, in't Veld B; European Society of Anaesthesiology. Perioperative fasting in adults and children: guidelines from the European Society of Anaesthesiology. Eur J Anaesthesiol. 2011 Aug;28(8):556-69. doi: 10.1097/EJA.0b013e3283495ba1. PMID 21712716
- [Background] Weimann A, Braga M, Carli F, Higashiguchi T, Hubner M, Klek S, Laviano A, Ljungqvist O, Lobo DN, Martindale R, Waitzberg DL, Bischoff SC, Singer P. ESPEN guideline: Clinical nutrition in surgery. Clin Nutr. 2017 Jun;36(3):623-650. doi: 10.1016/j.clnu.2017.02.013. Epub 2017 Mar 7. PMID 28385477
- [Background] Joshi GP, Abdelmalak BB, Weigel WA, Harbell MW, Kuo CI, Soriano SG, Stricker PA, Tipton T, Grant MD, Marbella AM, Agarkar M, Blanck JF, Domino KB. 2023 American Society of Anesthesiologists Practice Guidelines for Preoperative Fasting: Carbohydrate-containing Clear Liquids with or without Protein, Chewing Gum, and Pediatric Fasting Duration-A Modular Update of the 2017 American Society of Anesthesiologists Practice Guidelines for Preoperative Fasting. Anesthesiology. 2023 Feb 1;138(2):132-151. doi: 10.1097/ALN.0000000000004381. PMID 36629465
- [Background] Cheng PL, Loh EW, Chen JT, Tam KW. Effects of preoperative oral carbohydrate on postoperative discomfort in patients undergoing elective surgery: a meta-analysis of randomized controlled trials. Langenbecks Arch Surg. 2021 Jun;406(4):993-1005. doi: 10.1007/s00423-021-02110-2. Epub 2021 Feb 25. PMID 33629128
- [Background] Rizvanovic N, Nesek Adam V, Causevic S, Dervisevic S, Delibegovic S. A randomised controlled study of preoperative oral carbohydrate loading versus fasting in patients undergoing colorectal surgery. Int J Colorectal Dis. 2019 Sep;34(9):1551-1561. doi: 10.1007/s00384-019-03349-4. Epub 2019 Jul 15. PMID 31309323
- [Background] Liu B, Wang Y, Liu S, Zhao T, Zhao B, Jiang X, Ye L, Zhao L, Lv W, Zhang Y, Zheng T, Xue Y, Chen L, Chen L, Wu Y, Li Z, Yan J, Wang S, Sun X, Gao G, Qu Y, He S. A randomized controlled study of preoperative oral carbohydrate loading versus fasting in patients undergoing elective craniotomy. Clin Nutr. 2019 Oct;38(5):2106-2112. doi: 10.1016/j.clnu.2018.11.008. Epub 2018 Nov 17. PMID 30497695
- [Background] Nygren J. The metabolic effects of fasting and surgery. Best Pract Res Clin Anaesthesiol. 2006 Sep;20(3):429-38. doi: 10.1016/j.bpa.2006.02.004. PMID 17080694
- [Background] Nygren J, Thorell A, Jacobsson H, Larsson S, Schnell PO, Hylen L, Ljungqvist O. Preoperative gastric emptying. Effects of anxiety and oral carbohydrate administration. Ann Surg. 1995 Dec;222(6):728-34. doi: 10.1097/00000658-199512000-00006. PMID 8526579